CLINICAL TRIAL: NCT00804648
Title: Patient Satisfaction With Timolol Maleate in Sorbate, Generic Timolol Gel Forming Solution or Timolol Hemihydrate in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Patient Satisfaction With Timolol in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VPH0111
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma, Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- hemihydrate/maleate/maleate gel (Active Comparator): Period one - Timolol hemihydrate 0.5% Period two - Timolol maleate 0.5% Period three - Timolol maleate gel forming solution 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution
- maleate/maleate gel/hemihydrate (Active Comparator): Period one - Timolol maleate 0.5% Period two - Timolol maleate gel forming solution 0.5% Period three - Timolol hemihydrate 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution
- maleate gel/hemihydrate/maleate (Active Comparator): Period one - Timolol maleate gel forming solution 0.5% Period two - Timolol hemihydrate 0.5% Period three - Timolol maleate 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution
- hemihydrate/maleate gel/maleate (Active Comparator): Period one - Timolol hemihydrate 0.5% Period two - Timolol maleate gel forming solution 0.5% Period three - Timolol maleate 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution
- maleate/hemihydrate/maleate gel (Active Comparator): Period 1 - Timolol maleate 0.5% Period 2 - Timolol hemihydrate 0.5% Period 3 - Timolol maleate gel forming solution 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution
- maleate gel, maleate, hemihydrate (Active Comparator): Period 1 - Timolol maleate gel forming solution 0.5% Period 2 - Timolol maleate 0.5% Period 3 - Timolol hemihydrate 0.5%
  Interventions: Drug: Timolol Maleate in Sorbate; Drug: Timolol hemihydrate; Drug: Timolol maleate gel forming solution

INTERVENTIONS:
Drug: Timolol Maleate in Sorbate — 0.5%
Drug: Timolol hemihydrate — 0.5%
Drug: Timolol maleate gel forming solution — 0.5%

SUMMARY:
This study compares patient symptoms and anterior segment safety in patients treated with timolol hemihydrate, generic timolol gel forming solution or timolol maleate.

ELIGIBILITY:
Inclusion Criteria:

* willing to comply with investigator's and protocol's instructions
* patients signature on the informed consent document
* primary open-angle glaucoma, pigment dispersion or exfoliation glaucoma, or ocular hypertension in at least one eye
* at screening intraocular pressure must be considered to be safe, in both eyes
* in non-qualifying eyes the intraocular pressure should be able to be controlled safely on no pharmacologic therapy or on study medicine alone
* currently treated with one glaucoma medication, untreated intraocular pressure of less than or equal to 28 mm Hg at visit 2 in both eyes

Exclusion Criteria:

* any abnormality preventing reliable applanation tonometry in either eye
* any opacity or subject uncooperativeness that restricts adequate examination of the ocular fundus or anterior chamber in either eye
* any concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye
* any history of allergic hypersensitivity or poor tolerance to any components of the preparations used in this trial
* females of childbearing potential not using reliable means of birth control
* pregnant or lactating females
* any clinically significant, serious, or severe medical or psychiatric condition
* participation (or current participation) in any investigational drug or device trial within 30 days prior to Visit 1
* severe prior visual acuity or field loss from any cause
* inability to understand the trial procedures, and thus inability to give informed consent
* progressive retinal or optic nerve disease apart from glaucoma
* serious systemic or ocular disease
* intraocular laser surgery within the past three months or corneal or intraocular conventional surgery within the past 6 months
* concurrent use of systemic corticosteroids, by IV, oral, dermal or topical ophthalmic route.
* subjects requiring tear replacement drops or allergy medications with sympathomimetics 24 hours prior to a scheduled study visit
* contraindication to beta-blocker usage including: reactive airway disease, uncontrolled heart failure, or second as well as third degree cardiac block, myasthenia gravis
* any subject the investigator believes will be at risk for glaucomatous progression by their participation in this trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — PRN Pharmacuetical Research Network, LLC
Locations (2):
- United States (2):
  - Bourbonnais, Illinois
  - Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Maleate Gel/Maleate/Hemihydrate: Period 1 - Timolol maleate gel forming solution 0.5% Period 2 - Timolol maleate 0.5% Period 3 - Timolol hemihydrate 0.5%
Period: First Intervention
Arm/Group | Hemihydrate/Maleate/Maleate Gel | Maleate/Maleate Gel/Hemihydrate | Maleate Gel/Hemihydrate/Maleate | Hemihydrate/Maleate Gel/Maleate | Maleate/Hemihydrate/Maleate Gel | Maleate Gel/Maleate/Hemihydrate
Started | 3 | 5 | 6 | 4 | 4 | 8
Completed | 3 | 5 | 6 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Hemihydrate/Maleate/Maleate Gel | Maleate/Maleate Gel/Hemihydrate | Maleate Gel/Hemihydrate/Maleate | Hemihydrate/Maleate Gel/Maleate | Maleate/Hemihydrate/Maleate Gel | Maleate Gel/Maleate/Hemihydrate
Started | 3 | 5 | 6 | 4 | 4 | 8
Completed | 3 | 5 | 6 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Invervention
Arm/Group | Hemihydrate/Maleate/Maleate Gel | Maleate/Maleate Gel/Hemihydrate | Maleate Gel/Hemihydrate/Maleate | Hemihydrate/Maleate Gel/Maleate | Maleate/Hemihydrate/Maleate Gel | Maleate Gel/Maleate/Hemihydrate
Started | 3 | 5 | 6 | 4 | 4 | 8
Completed | 3 | 5 | 6 | 4 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Stinging on Instillation
Description: Assessed from subject response to survey question asking about tolerability of medicine upon instillation, using a 0 through 7 scale, with 0=complete comfort and 7=worst pain imaginable.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale | 0.6 (1.0) | 1.0 (1.4) | 0.6 (1.0)

2. Secondary Outcome: Conjunctival Hyperemia
Description: Assessed by investigator using a slit lamp and a photographic grading scale. Photographs were graded: grade 0, grade 1, grade 2, grade 3. The higher the graded the worse the hyperemia.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale | 0.2 (0.5) | 0.4 (0.5) | 0.3 (0.5)

3. Secondary Outcome: Tear Film Break-up Time
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Seconds | 8.5 (6.1) | 7.7 (4.9) | 8.5 (5.7)

4. Secondary Outcome: Corneal Staining Grade
Description: Assessed by the investigator using a slit lamp and Oxford Scheme, grading 0,1,2,3,4,5. The higher the grade the worse the staining.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale | 1.2 (0.9) | 1.1 (0.9) | 1.0 (0.8)

5. Secondary Outcome: Corneal Staining Count
Description: Assessed by the investigator using a slit lamp, counting the number of spots.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Number of spots
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Number of spots | 10.5 (12.5) | 10.4 (13.4) | 8.3 (8.3)

6. Secondary Outcome: Intraoclular Pressure
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: mm of mercury
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
mm of mercury | 16.3 (3.1) | 16.2 (2.4) | 16.2 (2.2)

7. Secondary Outcome: Basic Schirmer's
Description: Schirmer's measures basic tear function. The higher the number, the less dry the eye.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: mm of moisture
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
mm of moisture | 17.7 (9.7) | 14.8 (7.3) | 15.4 (6.4)

8. Secondary Outcome: Conjunctival Staining - Nasal Grade
Description: Assessed by investigator using a slit lamp and the Oxford Scheme, grading 0,1,2,3,4,5 according to pictures provided. The higher the grade the worse the staining.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale | 1.2 (0.9) | 1.1 (1.0) | 1.3 (1.0)

9. Secondary Outcome: Conjunctival Staining - Nasal Count
Description: Assessed by investigator using slit lamp and counting number of spots.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: number of spots
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
number of spots | 11.0 (12.5) | 10.3 (15.7) | 12.9 (14.8)

10. Secondary Outcome: Conjunctival Staining - Temporal Grade
Description: Assessed by investigator using a slit lamp and Oxford Scheme, grading 0,1,2,3,4,5 according to pictures provided. The higher the grade the worse the staining.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
Units on a scale | 0.8 (0.6) | 0.7 (0.7) | 0.8 (0.7)

11. Secondary Outcome: Conjunctival Staining - Temporal Count
Description: Assessed by investigator using a slit lamp and counting number of spots.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: number of spots
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
number of spots | 4.7 (7.3) | 4.8 (8.6) | 5.3 (6.7)

12. Secondary Outcome: Visual Acuity
Description: The visual acuity score is a count of the number of letters the subject successfully read from the eye chart. The higher the score, the better the vision.
Time Frame: following 3 days of treatment
Measure: Mean (Standard Deviation); unit: number of letters
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Number analyzed (Participants) | 30 | 30 | 30
number of letters | 52.3 (5.6) | 52.5 (6.1) | 51.4 (5.8)

ADVERSE EVENTS:
Arm/Group | Timolol Hemihydrate 0.5% | Timolol Maleate 0.5% | Timolol Maleate Gel Forming Solution 0.5%
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 2/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Timolol Hemihydrate 0.5% (N=30) | Timolol Maleate 0.5% (N=30) | Timolol Maleate Gel Forming Solution 0.5% (N=30)
Tearing (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the PI will provide the Sponsor with at least 60 days for review of a manuscript. If requested in writing, the PI will withhold publication for up to an additional 60 days.